CLINICAL TRIAL: NCT02701933
Title: Effects of Ketamine on Eye Movements, Perception and Brain Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Ulrich Ettinger, Professor of Psychology, University of Bonn
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: #14-03-20
Record Dates: First submitted 2016-02-17; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Functional Neuroimaging
MeSH Terms: interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine-Saline (Other): Each participant receives both ketamine and placebo (saline) in randomised order in a repeated-measures design. In this arm, ketamine is administered on the first assessment and placebo (saline) is administered on the second assessment.
  Interventions: Drug: Ketamine; Drug: Saline
- Saline-Ketamine (Other): Each participant receives both ketamine and placebo (saline) in randomised order in a repeated-measures design. In this arm, placebo (saline) is administered on the first assessment and ketamine is administered on the second assessment.
  Interventions: Drug: Ketamine; Drug: Saline

INTERVENTIONS:
Drug: Ketamine — Racemic ketamine, intravenous, at a concentration of 10mg ketamine per 50ml infusion
  Other Names: Ketamin Ratiopharm
Drug: Saline — Saline, intravenous infusion
  Other Names: Kochsalzloesung

SUMMARY:
In this study, the investigators examine the effects of low-dose ketamine on different oculomotor, perceptual and cognitive functions. They also examine effects on concurrent brain activity using blood oxygen level dependent (BOLD) functional magnetic resonance imaging (fMRI). A sample of N=25 healthy, male participants is required to complete the study. The design is within-subjects, placebo-controlled, double-blind and cross-over. A targeted ketamine level in plasma of 100ng/ml is applied. It is hypothesised that ketamine, compared to placebo, will lead to changes in task performance and brain activity similar to those observed in patients with schizophrenia.

DETAILED DESCRIPTION:
The uncompetitive N-methyl-D-aspartate (NMDA) receptor antagonist ketamine has been proposed as a model system of the symptoms of schizophrenia. To complement this model system and to allow neurobiological as well as translational studies, biomarkers are often applied to people under the influence of ketamine. Here, we apply oculomotor, perceptual and cognitive biomarkers to healthy human volunteers whilst they undergo BOLD fMRI at 3 Tesla field strength. We use a counter-balanced, placebo-controlled, double-blind, within-subjects design. A sample of 25 healthy participants is required. Participants will receive intravenous (IV) racemic ketamine (with a 100ng/ml target plasma concentration) on one of two assessment days and they will receive placebo (intravenous saline) on the other assessment day. BOLD fMRI will be carried out on a Siemens Trio scanner at the Life&Brain Centre, Bonn. In addition to brain functional and cognitive, perceptual and oculomotor responses, we will also measure self-ratings of psychosis-like experiences. These will be obtained using the Psychotomimetic States Inventory (PSI; Mason et al 2008).

ELIGIBILITY:
Inclusion Criteria:

* MRI-suitability
* suitability for video-based combined pupil and corneal reflection (VCPCR) eye-tracking
* good command of German language
* willingness to take part

Exclusion Criteria:

* any current or history of axis I disorder diagnosis as assessed by the Mini-International Neuropsychiatric Interview (M.I.N.I.)
* any neurological conditions and heart conditions
* use of any prescription or non-prescription medication up to one week before participation
* personal history of head-injuries, loss of consciousness, eye surgery or impairment of vision (other than corrective lenses)
* any other relevant medical conditions such as high blood pressure
* positive urine drug test (Drug-Screen Multi "5T", nal von minden GmbH)
* history of drug use or current drug use
* under- or overweight (below 18.5 and above 24.9 body mass index (BMI) values)
* any diagnosis of psychotic disorders among first-degree relatives

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Brain activity in cortical and subcortical areas as assessed using BOLD (blood oxygen level dependent) functional magnetic resonance imaging (fMRI) at 3 Tesla field strength | within 1 hour of start of IV infusion

SECONDARY OUTCOMES:
Psychotomimetic State Inventory (PSI) | within 1 hour of start of IV infusion
Visual Analogue Rating Scales (VARS) from Norris 1971; self-rating scores of the subscales "mental sedation", "physical sedation", "tranquillisation" and "other feelings and attitudes" | within 1 hour of start of IV infusion
d2 Attention Test, a measure of sustained attention | within 1 hour of start of IV infusion
  The test requires the crossing out of the letter d combined with two dashes amidst letters d and p combined with one, two, three or four dashes and is a well-established measure of sustained attention
Recognition memory performance (latencies in ms) | after 5 days of washout period
Recognition memory performance (percent correct responses) | after 5 days of washout period
Smooth pursuit gain (%) | within 1 hour of start of IV infusion
Smooth pursuit root mean square error (RMSE) | within 1 hour of start of IV infusion
Smooth pursuit saccadic frequency (number per second) | within 1 hour of start of IV infusion
Prosaccade latency (ms) | within 1 hour of start of IV infusion
Prosaccade gain (%) | within 1 hour of start of IV infusion
Prosaccade spatial error (%) | within 1 hour of start of IV infusion
Prosaccade velocity (degrees per second) | within 1 hour of start of IV infusion
Prosaccade error rate (%) | within 1 hour of start of IV infusion
Antisaccade latency (ms) | within 1 hour of start of IV infusion
Antisaccade gain (%) | within 1 hour of start of IV infusion
Antisaccade spatial error (%) | within 1 hour of start of IV infusion
Antisaccade velocity (degrees per second) | within 1 hour of start of IV infusion
Antisaccade error rate (%) | within 1 hour of start of IV infusion

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Ettinger, PhD, Principal Investigator — Department of Psychology, University of Bonn
Locations (1):
- University of Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No